CLINICAL TRIAL: NCT01225809
Title: Observational Follow-up Extension Study-visit to Evaluate Long-term Safety and Tolerability of Immunization With AFFITOPE AD01 Applied During AFFiRiS001 in Patients With Alzheimer's Disease
Brief Title: AD01 Follow up Extension Visit
Status: Completed | Type: Observational
Sponsor: Affiris AG (Industry)
Responsible Party: Achim Schneeberger; CMO, AFFiRiS AG
Other Study IDs: AFF003E
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer´s Disease
Keywords: AD01 follow-up extension

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AD01with or without adjuvant: Patients who have received at least one immunization of AD01 with or without adjuvant during AFF001

SUMMARY:
Patients who were vaccinated with AFFITOPE AD01 during AFFiRiS001 will undergo a long-term follow-up period to get more information regarding the safety profile of AFFITOPE AD01.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated by the patient or the patient's legal representative and the caregiver.
* Patients having participated in AFFiRiS 001 and AFF003 and having received ≥1 vaccination with AFFITOPE AD01
* Availability of a partner/caregiver knowing the patient

Exclusion Criteria:

* Patients having received no vaccination with AFFITOPE AD01
* History of questionable compliance to visit schedule

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having participated in AFFiRiS 001 and AFF003 and having received ≥1 vaccination with AFFITOPE AD01
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Long term tolerability and safety of AFFITOPE AD01 | One year.
  retrospective assessment of safety data

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dal-Bianco, MD, Principal Investigator — Univ. Klinik für Neurologie
Locations (1):
- Univ. Klinik für Neurologie, Vienna, Austria